CLINICAL TRIAL: NCT02013596
Title: Effect of Transcutaneous Electrical Acupoint Stimulation(TEAS) on the Hepatic and Renal Function Impaired by Pneumoperitoneum: a Prospective, Randomized Controlled Trial
Brief Title: Transcutaneous Electrical Acupoint Stimulation(TEAS) for Hepatic and Renal Dysfunction After Pneumoperitoneum
Acronym: TRIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhihong LU (Other)
Responsible Party: Sponsor-Investigator, Zhihong LU, Dr., Air Force Military Medical University, China
Organization: Air Force Military Medical University, China (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XJH-A-2013-08-2
Record Dates: First submitted 2013-09-16; First posted 2013-12-17 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2016-01

CONDITIONS: Hepatic Dysfunction Transient; Renal Function Disorder
Keywords: hepatic dysfunction; renal dysfunction; pneumoperitoneum; Transcutaneous electric stimulation
MeSH Terms: conditions — Liver Diseases; Renal Insufficiency; Pneumoperitoneum

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (No Intervention): Patients were given no TEAS
- TEAS Pretreatment (Experimental): Patients were given 30min of TEAS before pneumoperitoneum
  Interventions: Other: TEAS pretreatment
- TEAS Treatment (Experimental): Patients were given 30min of TEAS during pneumoperitoneum
  Interventions: Other: TEAS treatment

INTERVENTIONS:
Other: TEAS pretreatment — Electric stimulation was given through electrode attached to specific acupoints for 30mins before anesthesia induction
  Arms: TEAS Pretreatment
Other: TEAS treatment — Transcutaneous Electrical Acupoint Stimulation was given to the patient at the same time of the start of anesthesia induction for 30mins
  Arms: TEAS Treatment

SUMMARY:
The purpose of this study is to compare the effect of TEAS pretreatment and treatment on hepatic and renal dysfunction induced by pneumoperitoneum in patients undergoing laparoscopic surgeries.

DETAILED DESCRIPTION:
Patients were randomly assigned to three groups, control group and two intervention groups, receiving TEAS before and after general anesthesia induction respectively. TEAS was given through electrodes attached to acupoints. The time for TEAS was 30min. Venous blood samples were collected before and 20min after pneumoperitoneum. Hepatic and renal function index including AST, ALT, ALP, BUN, Cr were measured.

ELIGIBILITY:
Inclusion Criteria:

* Age>18yrs,<60yrs；
* ASA 1-2；
* Scheduled for laparoscopic surgery under general anesthesia；
* Informed consented

Exclusion Criteria:

* Patients with hepatic or renal dysfunction；
* Patients with severe hypertension or cardiac dysfunction；
* Patients with severe pulmonary disease；
* Patients with hemoglobin<100g/L

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 168 (Actual)
Dates: Start 2013-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Incidence of renal or hepatic dysfunction | 20min after pneumoperitoneum
  percentage of patients with renal or hepatic dysfunction

SECONDARY OUTCOMES:
Change of hepatic function | 20min after pneumoperitoneum
  the increase of hepatic ALT and AST after pneumoperitoneum
Change of renal function | 20min after pneumoperitoneum
  Change of BUN and Cr after pneumoperitoneum

CONTACTS AND LOCATIONS:
Overall Officials: zhihong Lu, MD, Principal Investigator — Air Force Military Medical University, China
Locations (1):
- Xijing Hospital, Fourth Military Medical University, Xi'an, Shaanxi, China

REFERENCES:
- [Background] Westgarth-Taylor C, de Lijster L, van Bogerijen G, Millar AJ, Karpelowsky J. A prospective assessment of renal oxygenation in children undergoing laparoscopy using near-infrared spectroscopy. Surg Endosc. 2013 Oct;27(10):3696-704. doi: 10.1007/s00464-013-2950-3. Epub 2013 Apr 19. PMID 23605192
- [Background] de Barros RF, Miranda ML, de Mattos AC, Gontijo JA, Silva VR, Iorio B, Bustorff-Silva JM. Kidney safety during surgical pneumoperitoneum: an experimental study in rats. Surg Endosc. 2012 Nov;26(11):3195-200. doi: 10.1007/s00464-012-2322-4. Epub 2012 May 19. PMID 22609982
- [Background] Parikh BK, Shah VR, Modi PR, Butala BP, Parikh GP. Anaesthesia for laparoscopic kidney transplantation: Influence of Trendelenburg position and CO2 pneumoperitoneum on cardiovascular, respiratory and renal function. Indian J Anaesth. 2013 May;57(3):253-8. doi: 10.4103/0019-5049.115607. PMID 23983283
- [Background] Wiesenthal JD, Fazio LM, Perks AE, Blew BD, Mazer D, Hare G, Honey RJ, Pace KT. Effect of pneumoperitoneum on renal tissue oxygenation and blood flow in a rat model. Urology. 2011 Jun;77(6):1508.e9-15. doi: 10.1016/j.urology.2011.02.022. Epub 2011 Apr 19. PMID 21507469
- [Background] Ahn JH, Lim CH, Chung HI, Choi SU, Youn SZ, Lim HJ. Postoperative renal function in patients is unaltered after robotic-assisted radical prostatectomy. Korean J Anesthesiol. 2011 Mar;60(3):192-7. doi: 10.4097/kjae.2011.60.3.192. Epub 2011 Mar 30. PMID 21490821
- [Background] Hoekstra LT, Ruys AT, Milstein DM, van Samkar G, van Berge Henegouwen MI, Heger M, Verheij J, van Gulik TM. Effects of prolonged pneumoperitoneum on hepatic perfusion during laparoscopy. Ann Surg. 2013 Feb;257(2):302-7. doi: 10.1097/SLA.0b013e31825d5b2b. PMID 22824851
- [Background] Eryilmaz HB, Memis D, Sezer A, Inal MT. The effects of different insufflation pressures on liver functions assessed with LiMON on patients undergoing laparoscopic cholecystectomy. ScientificWorldJournal. 2012;2012:172575. doi: 10.1100/2012/172575. Epub 2012 Apr 24. PMID 22619616
- [Background] Li J, Liu YH, Ye ZY, Liu HN, Ou S, Tian FZ. Two clinically relevant pressures of carbon dioxide pneumoperitoneum cause hepatic injury in a rabbit model. World J Gastroenterol. 2011 Aug 21;17(31):3652-8. doi: 10.3748/wjg.v17.i31.3652. PMID 21987614
- [Background] Jeong GA, Cho GS, Shin EJ, Lee MS, Kim HC, Song OP. Liver function alterations after laparoscopy-assisted gastrectomy for gastric cancer and its clinical significance. World J Gastroenterol. 2011 Jan 21;17(3):372-8. doi: 10.3748/wjg.v17.i3.372. PMID 21253398